CLINICAL TRIAL: NCT02035969
Title: A Randomized Controlled Trial to Assess the Effect of Group Peer Support to Children With HIV in Relation to Adherence, Virological Treatment Failure as Well as Physical Development
Brief Title: Assessment of Group Peer Support to Children With HIV in Vietnam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Mattias Larsson, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: K2012-56X-22028-01-3
Record Dates: First submitted 2013-12-17; First posted 2014-01-14 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment (CT) (No Intervention): Treatment according to the National Treatment Guidelines in Vietnam including treatment counseling and clinical follow up every three months. The caretaker of the child is responsible that the child will take the drugs and is provided with a pre-packed dosage form for easy remembering
- Enhanced Treatment Support (ETS) (Experimental): Treatment according to the National Treatment Guidelines in Vietnam including treatment counselling and clinical follow up every three months. In addition adherence support is provided according to the description under intervention.
  Interventions: Behavioral: Enhanced Treatment Support (ETS)

INTERVENTIONS:
Behavioral: Enhanced Treatment Support (ETS) — Peer supporters, who are also caregivers of HIV-infected children, organize peer support group meetings. In the meetings one peer supporter discusses problems related to adherence with caretakers and provides them with information. Another supporter provides children above 3 years of age with age relevant information about their disease and treatment as well as games and play to enhance group bounds. The supporter will also have weekly telephone contact with all caretakers to assess the condition of the child.
  For children with poor adherence individual support to caretakers and patients will be arranged to assess the child's condition and reason for poor adherence, in case of complications the supporter gives advice or refers the child for medical checkup.
  Arms: Enhanced Treatment Support (ETS)

SUMMARY:
This project aims to assess the effect of group peer support to children with HIV in relation to adherence, virological treatment failure as well as physical development. A randomised controlled trial (RCT) will be used where HIV+ children on antiretroviral treatment (ARV) and their caretakers are randomized into either enhanced treatment support (ETS) through peer supporters or the conventional treatment (CT) according to the guidelines of The National AIDS Control Program. The treatment strategies will be assessed and compared in relation to virological treatment failure as primary endpoint, immunological and clinical (AIDS events and mortality) as secondary endpoints as well as treatment adherence and physical development. The results from this project will lead to an increased knowledge in relation to the impact of enhanced treatment support on adherence, virological suppression and resistance development for children with HIV and have an impact on HIV treatment policies and guidelines for Pediatric HIV in low-income settings globally.

DETAILED DESCRIPTION:
Main Aim To study the impact of peer support to children with HIV on antiretroviral treatment (ART) in relation to adherence, virological treatment failure, HIV drug resistance development as well as physical development using a randomised controlled trial (RCT) design comparing enhanced treatment support (ETS) and conventional treatment (CT).

Specific Aims

1. To assess the rate and risk factors for virological treatment failure among children on ART for more than 6 months using HIV viral load in blood in relation to clinical and socioeconomic indicators.
2. To recruit 520 HIV+ children 0-12 years of age on ART and randomize to either enhanced treatment support (ETS) or conventional treatment (CT).
3. To monitor ART adherence, CD4+ T-cell count, HIV viral load, clinical status, physical and cognitive development AIDS-associated events and/or mortality during every 6 months during a 36 months follow up period.
4. To assess the effect of ETS compared to CT with respect to the primary endpoint, virological treatment failure and specific ART mutations as well as the secondary endpoints, immunological failure, ART adherence, physical and cognitive development, and mortality and/or AIDS events.
5. To conduct a cost effectiveness assessment comparing ETS and CT.

This is a multi center study that includes the National Pediatric Hospital in Hanoi and the two major pediatric hospitals in Ho Chi Minh City. A study population of 520 HIV+ children receiving ARTs will be recruited from these hospitals. The reason for selecting children on ART is to see if treatment support can be initiated successfully after initiation of ART. Each HIV+ patient is examined according to WHO guidelines. HIV+ children will receive a complete physical examination including clinical staging of HIV infection, opportunistic infections and evidence of tuberculosis. Laboratory testing will include full blood count, CD4+ T-cell count (for children under five years of age CD4 %), viral load using ExaVirR viral load and liver enzymes. If indicated (e.g. prolonged cough and/or fever) chest X-ray, sputum microscopy for AFB will be done.

Opportunistic infections in HIV+ patients will be treated according to national guidelines. HIV+ children and their caregivers receive counselling and clinical follow ups. Tuberculosis (TB) will be managed in collaboration with the National Tuberculosis Program.

Inclusion and exclusion criteria's are described below. The patients recruited will be stratified according to age, sex and identified risk factor, then they will be randomised into two different treatment strategies a) Enhanced treatment support (ETS) strategy (described below) and Conventional treatment (CT). The patients treated under the two strategies will be compared with respect to: (i) virological treatment failure, (ii) patient's adherence to treatment strategy, (iii) physical development, and (iv) mortality and AIDS event. First drug regimen for all patients includes stavudine or AZT, lamivudine, nevirapine or efavirens. All procedures, treatment, and follow up for adverse effects are done according to national guidelines. The health care workers are trained in regular monitoring of patients and implementation of optimal treatment strategy. All procedures and treatment will follow the national guidelines. Follow up visits including physical examinations, adherence evaluation and laboratory tests will be done every 3 months.

The tests will include full blood count and liver enzymes as well as other indicated tests. Viral load and CD4+ T-cell count will be monitored every 6 months.

The number of patients needed for each arm of the experiment was estimated assuming an absolute 2-year risk of treatment failure of 15% in the control arm. Assuming proportional hazards there is an absolute 2-year risk of failure in the peer-support group of 7%. Requiring a power of 80% and a significance level of 5% approximately 480 patients are required. In order to account for some losses to follow-up and deviations from our assumptions, we will recruit a total of 260 patients into each arm.

In the ETC strategy caretakers and children with HIV on ART will be supported to achieve better adherence through peer support groups at the beginning of treatment and phone follow-up later, with an option for home visits or to return to support groups later if necessary. The activities will be organized by peer supporters, caregivers of HIV-infected children selected by peers, who will undergo a series of training, including medication adherence and counselling skills. They will ideally be assigned to patients living in the same community or in proximity to patients in the intervention group.

Peer group meetings with 7-10 caretakers and children will be organized monthly according to age groups, e.g. 0-3 years, 4-6 years, 7-12 years, and location. In these meetings caretakers will discuss problems related to adherence and receive new information from peer supporters. Simultaneously, children above 3 years of age will receive age relevant information about their disease and treatment from another supporter as well as do games and play to enhance group bounds. The supporters will also have weekly telephone contact with the caretakers, if needed more, to assess the condition of the child. To those who cannot make a particular meeting or answer the phone home visits (if consent is given) are made. Follow up phone calls will be made to those whom the case manager identifies to need more support.

As children differ very much depending on age the intervention will be adjusted to each age group in order to provide the best possible support according to standardized procedures that can be replicated. For children with poor adherence individual support to caretakers and patients will be arranged where the condition of the child and reason for poor adherence is assessed, in case of complications the peer supporter will provide advice and if needed refer the child for medical checkup. In CT control group the treatment will be supported according to the treatment guidelines. Both groups will receive treatment counseling and be followed through regular clinical check-up, the drugs will be provided in a pre-packed dosage form for easy remembering and counting of the pills.

The patients are followed for 36 months and monitored each six months through viral load in plasma using ExaVir Load®, CD4+ T-cell count, adherence, clinical examination including physical development. Viral load will be assessed using a new ELISA based technique ExaVir Load® that detects HIV reverse transcriptase down to 1 fg/ml blood-plasma corresponding to 200 HIV RNA copies/ml. Adherence will be assessed every three months using questionnaires designed specifically for age groups. For infants and young children the Pediatric International Adherence Questionnaire (PIAQ) may be used, and for older children the Adult AIDS Clinical Trials Group (ACTG) Adherence Instruments will be used. The questionnaire interviews will be conducted by health personnel at the Out Patient Clinics for Pediatric HIV. Adherence will also be measured by pill count, where the patients bring their remaining drugs back to the clinic at follow-up, enabling calculation of the proportion of drugs remaining out of the total amount of prescribed drugs as well as through pharmacy records if the patients have collected the drugs accurately. Assessment of side effects will be done according to WHO suggested monitoring and management of ARV drugs together with the clinical examination each three months.

The primary endpoint will be virological treatment failure defined as a viral load corresponding to 1000 copies/ml. This could also be expressed as loss of virological response taking death and Loss of Follow Up into account. The secondary endpoints immunological treatment failure (no rise in CD4+ T-cell count at 1 year or decrease with 50% compared to the highest value or CD4+ T-cell count below 100), clinical treatment failure as defined by a new AIDS-defining illness or death due to HIV/AIDS (including TB and opportunistic infection) after starting treatment, and physiological development.

Costing of the two different strategies will be carried out by collecting monetary data of expense for drugs, test, allowance and other expenses from perspective of the HIV/AIDS treatment provider during ART. The investigators follow the basic principles of activity-based costing by identifying all activites necessary to provide the ETS and CT and then calculate the costs of carrying out each activity. Costs for each activity comprise recurrent and capital costs, direct and indirect costs. Recurrent costs are the routine costs of resources that are consumed within a year, i.e., non-capital items such as labor and medical supplies. Capital costs represent the annual portion of the cost of durable HIV Sida DOTARV assets. Effectiveness will be measured by percentages of patients with virological treatment failure defined as Viral Load >400 copise/ml.

The statistical analysis mainly consists in the comparison between the two groups with respect to the defined primary and secondary endpoints in relation to the semi-quantitative assessments of adherence. Standard statistical methods will be used. Hazard/Survival analysis will be conducted including death/loss of follow up as 'failure' in the analysis. Intention to treat will be used for analysis. Regression models with outcome as the dependent variable and a group indicator together with patient characteristics as independent variables will be the main approach. For binary outcomes, logistic regression will be used. Attention has to be paid to the particular, often skewed, distributions of variables like CD4+ T-cell counts and viral load. Transformations or the use of non-parametric approaches are likely to be necessary if such measures are not dichotomized and used in linear regression. The correlation between drug resistance and adherence will be statistically analyzed in order to study whether the basic mechanisms of selective drug pressure result in a concave or bell-shaped resistance - adherence relationship, for these drugs during ETS or CT in a low-income setting. The odds ratios of having or not baseline drug resistance mutations as detected by population and deep (single allele PCR) sequencing on drug resistance development and clinical outcomes during treatment independent of treatment adherence will be evaluated. Stratified analysis will be conducted comparing the outcomes among the treatment groups.

The investigators will strictly comply with widely recognized international texts and codes of practice including the Helsinki agreement. In this project one patient cohort will receive ETS and the other CT. However both groups will be encouraged to proceed regularly with their drug treatment and to present difficulties that they may encounter in doing so. For the project period, the project will meet the costs of ART for the cohorts. Patients' biological samples will be collected and used only after written consent from the children's caretaker. All specimens will be coded to protect the identity of patients and to ensure confidentiality. Patients will be recruited in a consecutive manner without regard to race or other exclusion considerations. Confidentiality will be assured by using codes for patient identification, and confidentially laws will be strictly observed when processing human clinical information. No patient identifying information will be published or available after the requisite clinical data has been collected, and consent will be obtained for the use of all data and tissues. Data will be accessible only to members and coordinators of the tissue procurement facility and research team, under approved guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Children already on first line ART

Exclusion Criteria:

* Children age above 12 years
* Children with institutionalized parents
* Children whose sibling are already included

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Estimated)
Dates: Start 2013-12; Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-04 (Estimated)

PRIMARY OUTCOMES:
Virological treatment failure | 24 months
  HIV viral load of 1000 copies/ml

SECONDARY OUTCOMES:
Immunological treatment failure | 24 months
  * No rise in CD4+ T-cell count after 1 year of treatment
  * 50% decline compared to the highest value
  * CD4+ T-cell count below 100

OTHER OUTCOMES:
Clinical treatment failure | 24 months
  Occurence or recurrence of stage 4 diseases or conditions after at least 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Larsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam